CLINICAL TRIAL: NCT02758002
Title: Inhibition of Atrial Fibrillation by Elimination of Transitional Mechanisms
Acronym: TRANS AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 151850
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: atrial fibrillation ablation; ablation; atrial fibrillation rotors
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Firm ablation for transitional AF rotors (Experimental): All subjects will undergo this ablation, in addition to their standard PVI and Firm ablation for sustained AF rotors.
  Interventions: Procedure: Firm ablation for transitional AF rotors

INTERVENTIONS:
Procedure: Firm ablation for transitional AF rotors — Transitional AF rotors will be mapped and ablated as part of this study. All subjects will undergo this ablation after standard PVI and Firm ablation for sustained rotors.

SUMMARY:
There is growing awareness of the importance of electrical rotors to the maintenance of atrial fibrillation (AF). Recent work in our laboratory has found that AF evolves over time, from rapid, focal activation, next to transitional rotors, and finally to stable, long duration rotors, whose locations are frequently separate from the transitional rotor sites. This project will test the hypothesis that mapping and ablation of the transitional rotors sites may prevent atrial fibrillation from progressing to sustained atrial fibrillation, and therefore increase the AF initiation threshold. The investigators will test this hypothesis during clinically-indicated electrophysiology study prior to ablation of symptomatic AF.

DETAILED DESCRIPTION:
A. Patient Enrollment:

UCSD will enroll subjects with symptomatic AF undergoing clinically-indicated ablation at the Sulpizio Cardiovascular Center.

B. Research Study Data UCSD will record patient demographics (e.g. age, gender, echocardiographic information), AF history (AF duration, previous and current antiarrhythmic medications, prior ablations), medical history (current medication regimen, lab values, etc.), and other relevant history. All recorded digital data such as electrocardiograms and intracardiac recordings will be exported from the recorder stripped of patient identifying information.

C. Electrophysiology (EP) Study and Catheter Placement:

EP study will be performed in the fasting state and after antiarrhythmic medications are discontinued for 5 half-lives (>60 days for amiodarone). Catheters are advanced to the right atrium (RA), coronary sinus, and transseptally to left atrium (LA). A 64-pole basket catheter (FIRMap, Topera, Menlo Park, CA) will map the LA. RA recordings are made using a second basket, simultaneously when possible. Heparin will be infused to maintain activated clotting time >350 seconds.

D. Data Acquisition:

Creating an Electroanatomic Map Digital electroanatomical maps ("shells") will be created of each atrium's using mapping software (Ensite NavX, St Jude, St. Paul, MN or Biosense-Webster, Carto, Diamond Bar, CA.) Each shell is created by sampling atrial and venous points (Figure 3), and when available, referenced to preprocedural computed tomographic scans.

Recording Electrograms All AF electrograms will be recorded in a wide field-of-view using the 64-pole basket catheters. Unipolar and bipolar electrograms are filtered at 0.05 Hz to 500 Hz and recorded at 1 kHz (Bard, Lowell, MA) as described in prior work9.

Inducing AF Induction will be performed systematically first with programmed premature atrial contractions (PACs) using single extrastimuli at shortening coupling intervals after an 8-beat drive of cycle length (CL) 500ms (120 bpm). Next, burst pacing will be done at CL 500ms, reducing in 50ms steps to 300ms, then in 10ms steps to AF from the proximal coronary sinus as a stable reference point. If AF still does not initiate, isoproterenol (≤ 10mcg/min)10 will be infused. Each patient's induction threshold will be documented.

Recording Transitional and Sustained AF AF from induction until >5 minutes will be recorded, at which point prior work suggests AF is sustained, 6 whether spontaneous or induced. The first few seconds of AF will then be analyzed as described below.

9.2 Data Analysis A. AF initiation will be mapped and transitional mechanisms identified Phase mapping will be used to analyze AF initiation, defined as the first 5 seconds of AF. Biatrial phase movies will be created to visualize spatial distribution of activation times across the LA and RA. These phase movies illustrate the rotor phase singularities, which are defined as the point about which the integral of phase is 0, and visualized as the intersection of depolarization and repolarization isolines.

In patients with multiple AF initiations, the investigators will determine whether AF initiation occurs at conserved sites, defined as a separation in location ≤1 electrode distance. Other initiating mechanisms will be noted, including rapidly-firing focal impulses (focal activation is defined as centrifugal emanation from an origin that drives the atrium into fibrillatory conduction.)

B. Transitional rotors will be ablated After identifying transitional AF rotors, they will be targeted for localized ablation. Rotor location within the atria will be noted, both in the electroanatomic map and relative to the basket catheter splines. Radiofrequency (RF) energy will be applied to the core of the rotor, as described previously6, 9. RF energy will be delivered with a 3.5 mm tip irrigated catheter (ThermoCool, Biosense-Webster) at 25-35 W or, in patients with heart failure, an 8 mm tip catheter (Blazer, Boston Scientific, Marlborough, MA) at 50 to 55 W, with a target temperature of 52˚C. Each lesion is applied for approximately 30-60 seconds, with a predetermined goal of 5-10 minutes of RF energy being placed to cover the ≈2 cm2 area of AF rotor precession.

C. Induction thresholds will be compared Post-ablation, AF will again be induced systematically using the same protocol as before, and this threshold will be compared to the pre-ablation one. The threshold will be considered as increased if the post-ablation induction protocol entails a more aggressive pacing protocol (e.g. a protocol with faster pacing [shorter cycle length]). Figure 4 summarizes the workflow for Specific Aim 2.

D. Sustained AF will be mapped and ablated FIRM maps of ongoing AF will be created and analyzed using RhythmView (Topera, Menlo Park, CA). Rotors and focal impulses are considered AF sources only if stable in repeated samples, to distinguish from transient fibrillatory activity. The focal source origin or rotor core (center of rotational activity) will be located by its electrode coordinates and localized digitally within each patient-specific anatomic shell at the time of each FIRM map to eliminate errors from subsequent possible movement.

Patients begin in sinus rhythm. If induction threshold is higher after ablating initiating mechanisms, rotor ablation will proceed as per standard. If induction threshold is not higher, AF initiation is re-mapped once to confirm elimination of initiating mechanism; if present, it will be ablated again and again re-mapped to confirm. DCCV: Direct-current cardioversion.

In this trial, the only aspects of the procedure that are specifically done for research are the mapping and ablating of the initiating rotors that are identified within the first minute of inducing AF. The mapping and ablating of the sustaining rotors and the following PVI ablation are all standard of care ablation procedures.

9.3 Study Follow-up Schedule

Enrolled subjects will be followed for 1 year in this study by one of the sub-investigators or the principle investigator. All study visits are considered standard of care and these clinic visits will be expected of patients that receive ablation, regardless of whether they enroll in the trial or not. This study will entail three in-clinic follow-up visits at 1month, 6month, and 12 months post-ablation. At these visits, the following information will be collected:

* Cardiovascular symptoms (such as shortness of breath, fatigue, palpitations)
* Physical exam
* Cardiac medications, including anti arrhythmics, and changes in prescriptions
* 12-lead ECG recordings
* Cardiac monitoring, including Holter monitor (of any duration) or event monitor (or any duration), should be reviewed for any arrhythmias. If present, implanted devices will be interrogated at this time, evaluating for the same.

A study visit window of +/- 2 weeks will be put into effect during study follow-up in order to better schedule and accommodate enrolled subjects' schedules.

9.4 Expected Results and Endpoints A. Ablation of transitional AF mechanisms will increase AF induction threshold. Preliminary work in the UCSD lab has found that ablation of a transitional rotor in a patient with paroxysmal AF increased the AF induction threshold. If this finding holds true for the proposed study, this will be an important mechanistic finding, of interest to the general electrophysiology community.

B. Ablation of transitional AF mechanisms will improve ablation success The secondary endpoint is 1-year survival free of AF, with follow-up as per guidelines (i.e. 24-hour Holter monitor every 6 months with 12-lead ECG at every follow-up visit.) The investigators expect ablation of transitional mechanisms will improve success versus historical controls matched by age, AF duration, LA size, and EF.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic atrial fibrillation (AF) undergoing clinically-indicated ablation
* either persistent or paroxysmal AF

Exclusion Criteria:

* decompensated heart failure;
* non-revascularized coronary ischemia
* LA diameter > 60mm
* inability or refusal to provide consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in AF threshold induction from ablation of transitional rotors | 1 day
  In patients presenting for AF ablation, the investigator will prospectively determine whether ablation of AF-initiating sites renders AF more difficult to induce, as measured by the rapid pacing cycle length required to initiate AF during two induction attempts consisting of rapid pacing of 15 seconds duration at decreasing cycle lengths.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Schricker, MD, MS, Principal Investigator — UCSD School of Medicine / San Diego Veteran's Affairs Hospital
Locations (1):
- Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schricker AA, Lalani GG, Krummen DE, Rappel WJ, Narayan SM. Human atrial fibrillation initiates via organized rather than disorganized mechanisms. Circ Arrhythm Electrophysiol. 2014 Oct;7(5):816-24. doi: 10.1161/CIRCEP.113.001289. Epub 2014 Sep 12. PMID 25217042
- [Background] Weerasooriya R, Khairy P, Litalien J, Macle L, Hocini M, Sacher F, Lellouche N, Knecht S, Wright M, Nault I, Miyazaki S, Scavee C, Clementy J, Haissaguerre M, Jais P. Catheter ablation for atrial fibrillation: are results maintained at 5 years of follow-up? J Am Coll Cardiol. 2011 Jan 11;57(2):160-6. doi: 10.1016/j.jacc.2010.05.061. PMID 21211687
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] Narayan SM, Baykaner T, Clopton P, Schricker A, Lalani GG, Krummen DE, Shivkumar K, Miller JM. Ablation of rotor and focal sources reduces late recurrence of atrial fibrillation compared with trigger ablation alone: extended follow-up of the CONFIRM trial (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation). J Am Coll Cardiol. 2014 May 6;63(17):1761-8. doi: 10.1016/j.jacc.2014.02.543. Epub 2014 Mar 13. PMID 24632280
- [Background] Miller JM, Kowal RC, Swarup V, Daubert JP, Daoud EG, Day JD, Ellenbogen KA, Hummel JD, Baykaner T, Krummen DE, Narayan SM, Reddy VY, Shivkumar K, Steinberg JS, Wheelan KR. Initial independent outcomes from focal impulse and rotor modulation ablation for atrial fibrillation: multicenter FIRM registry. J Cardiovasc Electrophysiol. 2014 Sep;25(9):921-929. doi: 10.1111/jce.12474. Epub 2014 Jul 23. PMID 24948520
- [Background] Narayan SM, Krummen DE, Rappel WJ. Clinical mapping approach to diagnose electrical rotors and focal impulse sources for human atrial fibrillation. J Cardiovasc Electrophysiol. 2012 May;23(5):447-54. doi: 10.1111/j.1540-8167.2012.02332.x. Epub 2012 Apr 26. PMID 22537106
- [Background] Chen SA, Hsieh MH, Tai CT, Tsai CF, Prakash VS, Yu WC, Hsu TL, Ding YA, Chang MS. Initiation of atrial fibrillation by ectopic beats originating from the pulmonary veins: electrophysiological characteristics, pharmacological responses, and effects of radiofrequency ablation. Circulation. 1999 Nov 2;100(18):1879-86. doi: 10.1161/01.cir.100.18.1879. PMID 10545432
- [Background] Oral H, Pappone C, Chugh A, Good E, Bogun F, Pelosi F Jr, Bates ER, Lehmann MH, Vicedomini G, Augello G, Agricola E, Sala S, Santinelli V, Morady F. Circumferential pulmonary-vein ablation for chronic atrial fibrillation. N Engl J Med. 2006 Mar 2;354(9):934-41. doi: 10.1056/NEJMoa050955. PMID 16510747
- [Background] Cosedis Nielsen J, Johannessen A, Raatikainen P, Hindricks G, Walfridsson H, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Hansen PS. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation. N Engl J Med. 2012 Oct 25;367(17):1587-95. doi: 10.1056/NEJMoa1113566. PMID 23094720
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Sommer P, Kircher S, Rolf S, John S, Arya A, Dinov B, Richter S, Bollmann A, Hindricks G. Successful Repeat Catheter Ablation of Recurrent Longstanding Persistent Atrial Fibrillation With Rotor Elimination as the Procedural Endpoint: A Case Series. J Cardiovasc Electrophysiol. 2016 Mar;27(3):274-80. doi: 10.1111/jce.12874. Epub 2015 Dec 21. PMID 26527103
- [Background] Orlov MV, Gorev MV, Griben A. Rotors of truly atypical atrial flutters visualized by FIRM mapping and 3D-MRI overlay on live fluoroscopy. J Interv Card Electrophysiol. 2013 Dec;38(3):167. doi: 10.1007/s10840-013-9828-0. Epub 2013 Sep 12. PMID 24026969
- [Background] Deshmukh A, Patel NJ, Pant S, Shah N, Chothani A, Mehta K, Grover P, Singh V, Vallurupalli S, Savani GT, Badheka A, Tuliani T, Dabhadkar K, Dibu G, Reddy YM, Sewani A, Kowalski M, Mitrani R, Paydak H, Viles-Gonzalez JF. In-hospital complications associated with catheter ablation of atrial fibrillation in the United States between 2000 and 2010: analysis of 93 801 procedures. Circulation. 2013 Nov 5;128(19):2104-12. doi: 10.1161/CIRCULATIONAHA.113.003862. Epub 2013 Sep 23. PMID 24061087
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] O'Neill MD, Wright M, Knecht S, Jais P, Hocini M, Takahashi Y, Jonsson A, Sacher F, Matsuo S, Lim KT, Arantes L, Derval N, Lellouche N, Nault I, Bordachar P, Clementy J, Haissaguerre M. Long-term follow-up of persistent atrial fibrillation ablation using termination as a procedural endpoint. Eur Heart J. 2009 May;30(9):1105-12. doi: 10.1093/eurheartj/ehp063. Epub 2009 Mar 8. PMID 19270341
- [Background] Elayi CS, Verma A, Di Biase L, Ching CK, Patel D, Barrett C, Martin D, Rong B, Fahmy TS, Khaykin Y, Hongo R, Hao S, Pelargonio G, Dello Russo A, Casella M, Santarelli P, Potenza D, Fanelli R, Massaro R, Arruda M, Schweikert RA, Natale A. Ablation for longstanding permanent atrial fibrillation: results from a randomized study comparing three different strategies. Heart Rhythm. 2008 Dec;5(12):1658-64. doi: 10.1016/j.hrthm.2008.09.016. Epub 2008 Sep 17. PMID 19084800
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Saksena S, Slee A, Waldo AL, Freemantle N, Reynolds M, Rosenberg Y, Rathod S, Grant S, Thomas E, Wyse DG. Cardiovascular outcomes in the AFFIRM Trial (Atrial Fibrillation Follow-Up Investigation of Rhythm Management). An assessment of individual antiarrhythmic drug therapies compared with rate control with propensity score-matched analyses. J Am Coll Cardiol. 2011 Nov 1;58(19):1975-85. doi: 10.1016/j.jacc.2011.07.036. PMID 22032709